CLINICAL TRIAL: NCT03992963
Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application
Brief Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application - 2019_04
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2019_04
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hearing Aid without frequency lowering enabled (Active Comparator)
  Interventions: Device: Hearing Aid without frequency lowering enabled
- Hearing Aid with frequency lowering enabled (Experimental)
  Interventions: Device: Hearing Aid with frequency lowering enabled

INTERVENTIONS:
Device: Hearing Aid without frequency lowering enabled — Each participant will be fitted with frequency lowering disabled. Disabled means standard hearing loss compensation without lowering higher frequencies in lower frequency areas. The input frequency is mapped to the same frequency in output.
  Arms: Hearing Aid without frequency lowering enabled
Device: Hearing Aid with frequency lowering enabled — Each participant will be fitted with frequency lowering enabled. The principle of the frequency lowering algorithm is to lower high frequencies to a lower frequency region with the aim of ensuring high frequency audibility to improve auditory emotion recognition.
  Arms: Hearing Aid with frequency lowering enabled

SUMMARY:
Participants will take part in both a passive and active emotion recognition task: (1) passively listening to semantically-neutral sentences with emotional prosody, and (2) actively listening and subsequently categorizing emotional sentences and sounds. Participants are seated and instructed to stare at a fixation cross while the stimulus is played. During this study, non-invasive physiological measurements of pupil dilation will be recorded from the participants. Using this paradigm we will be assessing the effect of frequency lowering on emotion recognition. The study takes the form of a partly three factorial design (passive task x frequency lowering x acclimatization). Participants also perform a two factor design (active task x frequency lowering). Each participant performs two passive tests (20 minutes long each) with frequency lowering on and off, and a four week acclimatization period in-between. Participants perform one active listening task after the acclimatization period with frequency lowering on and off.

ELIGIBILITY:
Inclusion Criteria:

* Healthy outer ear (without previous surgical procedures)
* Ability to fill in a questionnaire conscientiously
* Informed Consent as documented by signature
* Minimum 1 year hearing aid experience
* Moderate-Severe (N3-N5) hearing loss or Normal Hearing

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Known central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Changes in event-related-pupil-dilations (ERPDs) data | 6 weeks
  Pupil dilations will be recorded from the participant both before and during the performance of the auditory tasks. Analyses will be carried out relative to the baseline recording (made before the auditory tasks) and also the pre-trial baseline (measured one second prior to the onset of the stimulus), in order to account for differences in baseline physiological activity. It is planned to analyse event-related-pupil-dilations (ERPDs).

SECONDARY OUTCOMES:
self-perceived speech intelligibility rating | 6 weeks
  Subjective speech intelligibility will be assessed through self-perceived speech intelligibility on a continuous scale from 0 (nothing) to 100 (everything) during a training phase only.
behavioral emotion recognition categorical rating | 6 weeks
  Behavioral ratings will be assessed in the final stage of the study during the active task. Participants will categorize stimuli into emotion categories (happy, sad, etc.) in a forced-choice task after each auditory stimulus is played.
behavioral emotion recognition continuous rating | 6 weeks
  Behavioral ratings will be assessed in the final stage of the study during the active task. Participants rate the valence and arousal of the stimulus on a continuous scale from 1 (very low) to 9 (very high) after each auditory stimulus is played.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Raether, Principal Investigator — Sonova AG
Locations (1):
- Sonova AG, Stäfa, Switzerland

IPD SHARING:
Plan to Share IPD: No